CLINICAL TRIAL: NCT00973882
Title: Phase II Multicenter Study Evaluating the Efficacy of Carboplatin-Etoposide Combination in Hormone-resistant Prostate Cancers With Neuroendocrine Differentiation.
Brief Title: Carboplatin-Etoposide Combination in Hormone-Resistant Prostate Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARBETOP; ET2005-005
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Prostate Cancer
Keywords: Hormone resistant prostate cancer; Neuro-endocrine marker; Carboplatin-Etoposide combination; Neuro-endocrine differentiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin-Etoposide (Experimental)
  Interventions: Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC4 on day 1 repeated every 3 weeks for a maximum of 6 cycles
Drug: Etoposide — Etoposide 100 mg/m2 on day 1, day 2 and day 3 repeated every 3 weeks for a maximum of 6 cycles

SUMMARY:
The aim of our study is to assess the efficacy and toxicity of a chemotherapy regimen combining carboplatin and etoposide in patients with metastatic hormone-resistant prostate cancer and neuro-endocrine differentiation. Eligible patients are treated with the combination of carboplatin AUC4 on day 1 and etoposide 100 mg/m2 on day 1, day 2 and day 3 repeated every 3 weeks for a maximum of 6 cycles. Efficacy endpoints include Prostate Specific Antigen (PSA) and neuro-endocrine marker response (defined as a 50% or greater decrease from baseline serum values), objective response rate (according to RECIST criteria), and toxicity.

DETAILED DESCRIPTION:
Neuro-endocrine differentiation is observed in the evolution of hormone-resistant prostate cancer. The aim of our study is to assess the efficacy and toxicity of a chemotherapy regimen combining carboplatin and etoposide in patients with metastatic hormone-resistant prostate cancer and neuro-endocrine differentiation. To be eligible, patients must have either circulating neuro-endocrine markers (Chromogranin A: CgA, Neuron Specific Enolase: NSE)and/or visceral metastases. Eligible patients are treated with the combination of carboplatin AUC4 administered on day 1 and etoposide 100 mg/m2 given on day 1, day 2 and day 3 and repeated every 3 weeks for a maximum of 6 cycles. The primary objective of the study is to assess objective response to the carboplatin - etoposide combination (according to RECIST criteria for lesions and defined as a 50% or greater decrease from baseline serum values for PSA and neuro-endocrine markers). Secondary objectives include evaluation of toxicity, duration of response, progression-free-survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of prostate adenocarcinoma
* Metastatic disease, either measurable (lymph nodes, hepatic lesion, pulmonary lesions with longest diameter > or = 1 cm on spiral scan), or non measurable (bone metastasis)
* Patients must:

  * Have received hormonal therapy via surgical or chemical castration (LH-RH agonist) with or without anti-androgens. Anti-androgen withdrawal is recommended before inclusion, with an off-treatment period of at least 4 weeks. LH-RH agonist treatment must be continued.
  * Have a relapse or disease refractory to hormonal treatment (defined by a testosterone level < 0.5 µg/ml)
  * Have neuroendocrine progression defined, whatever the PSA level, as:

    * NSE and/or Chromogranin A > 1.5 x upper limit of normal (ULN) with or without visceral metastases (liver, lung, lymph node)
    * No increase of NSE or Chromogranin A, but visceral metastases (either hepatic, pleuro-pulmonary, or nodal) with cytological or histological confirmation of the presence of an undifferentiated or neuro-endocrine component of prostatic origin
* Prior treatment by radiotherapy is allowed but radiation therapy must have been completed for at least 4 weeks before inclusion and irradiated areas must not represent more than 25% of marrow reserves
* Prior treatment by estramustine is allowed but must have been stopped at least 4 weeks before inclusion
* Age> or = 18 years
* Life expectancy> or = 3 months
* Karnofsky index> or = 50%
* Adequate haematological function: neutrophils> or = 1.5 G/l, platelets> or = 100 G/l, haemoglobin> or = 8 g/dl. Use of erythropoietin is allowed.
* Adequate liver function: bilirubin level within the institution's normal range, AST and ALT< or = 1.5 ULN
* Adequate renal function: creatinine clearance> or = 40 ml/min (Gault and Cockroft method)
* Signed written informed consent.

Exclusion Criteria:

* Patients having no> 1.5 x ULN increase of at least one neuro-endocrine marker (NSE or chromogranin A) and no cytological or histological (undifferentiated or neuro-endocrine type) evidence of visceral metastasis (hepatic, pleuro-pulmonary, or nodal)
* History of other malignancies, other than curatively treated basal cell skin carcinoma or any other curatively treated cancer with no sign of recurrence within 5 years
* Symptomatically uncontrolled brain metastasis
* Interstitial radiation therapy (using strontium or samarium) within the previous 3 months
* Prior treatment with platinum salts or etoposide. Other chemotherapy regimens are allowed provided that the last dose has been administered> or = 4 weeks prior to inclusion.
* Concomitant treatment with other anti-cancer drugs, except corticoid or LH-RH agonist injections
* Peripheral neuropathy> or = 2 (NCI-CTCAE)
* Uncontrolled progressive thrombo-embolic disease
* Uncontrolled infection
* Medical history of acute myocardial infection or uncontrolled angina pectoris, or hypertension or uncontrolled arrythmia
* Inclusion in another clinical trial
* Impaired follow-up for social, geographical, familial or psychological reasons
* Any other unstable disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (clinical and/or biological): Clinical: objective response of target lesions according to RECIST criteria Biological: greater than 50% decrease of PSA, NSE and Chromogranin A levels | Every 6 weeks during treatment (6 cycles of carboplatin-etoposide) and 3 to 4 weeks after the end of treatment

SECONDARY OUTCOMES:
Duration of response (clinical and/or biological) | Every three months until progression
Toxicity | Every 3 weeks during treatment
Progression-free survival and overall survival | Every three months until progression

CONTACTS AND LOCATIONS:
Overall Officials: FLECHON Aude, MD, Principal Investigator — Centre Leon Berard
Locations (11):
- France (11):
  - Centre François Baclesse, Caen
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Institut Curie, Paris
  - Fondation Hôpital Saint-Joseph, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Background] Aumuller G, Leonhardt M, Janssen M, Konrad L, Bjartell A, Abrahamsson PA. Neurogenic origin of human prostate endocrine cells. Urology. 1999 May;53(5):1041-8. doi: 10.1016/s0090-4295(98)00631-1. PMID 10223503
- [Background] Bonkhoff H, Stein U, Remberger K. Endocrine-paracrine cell types in the prostate and prostatic adenocarcinoma are postmitotic cells. Hum Pathol. 1995 Feb;26(2):167-70. doi: 10.1016/0046-8177(95)90033-0. PMID 7532147
- [Background] Krijnen JL, Janssen PJ, Ruizeveld de Winter JA, van Krimpen H, Schroder FH, van der Kwast TH. Do neuroendocrine cells in human prostate cancer express androgen receptor? Histochemistry. 1993 Nov;100(5):393-8. doi: 10.1007/BF00268938. PMID 8307781
- [Background] Hansson J, Abrahamsson PA. Neuroendocrine pathogenesis in adenocarcinoma of the prostate. Ann Oncol. 2001;12 Suppl 2:S145-52. doi: 10.1093/annonc/12.suppl_2.s145. PMID 11762343
- [Background] Abrahamsson PA. Neuroendocrine differentiation in prostatic carcinoma. Prostate. 1999 May;39(2):135-48. doi: 10.1002/(sici)1097-0045(19990501)39:23.0.co;2-s. PMID 10221570
- [Background] Oesterling JE, Hauzeur CG, Farrow GM. Small cell anaplastic carcinoma of the prostate: a clinical, pathological and immunohistological study of 27 patients. J Urol. 1992 Mar;147(3 Pt 2):804-7. doi: 10.1016/s0022-5347(17)37390-1. PMID 1311395
- [Background] Kreis W. Current chemotherapy and future directions in research for the treatment of advanced hormone-refractory prostate cancer. Cancer Invest. 1995;13(3):296-312. doi: 10.3109/07357909509094465. No abstract available. PMID 7743383
- [Background] Tannock IF, Osoba D, Stockler MR, Ernst DS, Neville AJ, Moore MJ, Armitage GR, Wilson JJ, Venner PM, Coppin CM, Murphy KC. Chemotherapy with mitoxantrone plus prednisone or prednisone alone for symptomatic hormone-resistant prostate cancer: a Canadian randomized trial with palliative end points. J Clin Oncol. 1996 Jun;14(6):1756-64. doi: 10.1200/JCO.1996.14.6.1756. PMID 8656243
- [Background] Moore MJ, Osoba D, Murphy K, Tannock IF, Armitage A, Findlay B, Coppin C, Neville A, Venner P, Wilson J. Use of palliative end points to evaluate the effects of mitoxantrone and low-dose prednisone in patients with hormonally resistant prostate cancer. J Clin Oncol. 1994 Apr;12(4):689-94. doi: 10.1200/JCO.1994.12.4.689. PMID 7512127
- [Background] Calvert AH, Newell DR, Gumbrell LA, O'Reilly S, Burnell M, Boxall FE, Siddik ZH, Judson IR, Gore ME, Wiltshaw E. Carboplatin dosage: prospective evaluation of a simple formula based on renal function. J Clin Oncol. 1989 Nov;7(11):1748-56. doi: 10.1200/JCO.1989.7.11.1748. PMID 2681557
- [Background] Chatelut E, Canal P, Brunner V, Chevreau C, Pujol A, Boneu A, Roche H, Houin G, Bugat R. Prediction of carboplatin clearance from standard morphological and biological patient characteristics. J Natl Cancer Inst. 1995 Apr 19;87(8):573-80. doi: 10.1093/jnci/87.8.573. PMID 7752255
- [Background] Maksymiuk AW, Jett JR, Earle JD, Su JQ, Diegert FA, Mailliard JA, Kardinal CG, Krook JE, Veeder MH, Wiesenfeld M, et al. Sequencing and schedule effects of cisplatin plus etoposide in small-cell lung cancer: results of a North Central Cancer Treatment Group randomized clinical trial. J Clin Oncol. 1994 Jan;12(1):70-6. doi: 10.1200/JCO.1994.12.1.70. PMID 8270988
- [Background] Loehrer PJ Sr, Ansari R, Gonin R, Monaco F, Fisher W, Sandler A, Einhorn LH. Cisplatin plus etoposide with and without ifosfamide in extensive small-cell lung cancer: a Hoosier Oncology Group study. J Clin Oncol. 1995 Oct;13(10):2594-9. doi: 10.1200/JCO.1995.13.10.2594. PMID 7595712
- [Background] Miller AA, Herndon JE 2nd, Hollis DR, Ellerton J, Langleben A, Richards F 2nd, Green MR. Schedule dependency of 21-day oral versus 3-day intravenous etoposide in combination with intravenous cisplatin in extensive-stage small-cell lung cancer: a randomized phase III study of the Cancer and Leukemia Group B. J Clin Oncol. 1995 Aug;13(8):1871-9. doi: 10.1200/JCO.1995.13.8.1871. PMID 7636529
- [Background] Larive S, Bombaron P, Riou R, Fournel P, Perol M, Lena H, Dussopt C, Philip-Joet F, Touraine F, Lecaer H, Souquet PJ; Groupe Lyon-Saint Etienne d'Oncologie Thoracique. Carboplatin-etoposide combination in small cell lung cancer patients older than 70 years: a phase II trial. Lung Cancer. 2002 Jan;35(1):1-7. doi: 10.1016/s0169-5002(01)00288-4. PMID 11750705
- [Background] Okamoto H, Watanabe K, Nishiwaki Y, Mori K, Kurita Y, Hayashi I, Masutani M, Nakata K, Tsuchiya S, Isobe H, Saijo N. Phase II study of area under the plasma-concentration-versus-time curve-based carboplatin plus standard-dose intravenous etoposide in elderly patients with small-cell lung cancer. J Clin Oncol. 1999 Nov;17(11):3540-5. doi: 10.1200/JCO.1999.17.11.3540. PMID 10550152
- [Background] Quoix E, Breton JL, Daniel C, Jacoulet P, Debieuvre D, Paillot N, Kessler R, Moreau L, Coetmeur D, Lemarie E, Milleron B. Etoposide phosphate with carboplatin in the treatment of elderly patients with small-cell lung cancer: a phase II study. Ann Oncol. 2001 Jul;12(7):957-62. doi: 10.1023/a:1011171722175. PMID 11521802
- [Background] Papandreou CN, Daliani DD, Thall PF, Tu SM, Wang X, Reyes A, Troncoso P, Logothetis CJ. Results of a phase II study with doxorubicin, etoposide, and cisplatin in patients with fully characterized small-cell carcinoma of the prostate. J Clin Oncol. 2002 Jul 15;20(14):3072-80. doi: 10.1200/JCO.2002.12.065. PMID 12118020
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc 53:457-81, 1958
- [Result] Flechon A, Pouessel D, Ferlay C, Perol D, Beuzeboc P, Gravis G, Joly F, Oudard S, Deplanque G, Zanetta S, Fargeot P, Priou F, Droz JP, Culine S. Phase II study of carboplatin and etoposide in patients with anaplastic progressive metastatic castration-resistant prostate cancer (mCRPC) with or without neuroendocrine differentiation: results of the French Genito-Urinary Tumor Group (GETUG) P01 trial. Ann Oncol. 2011 Nov;22(11):2476-2481. doi: 10.1093/annonc/mdr004. Epub 2011 Mar 24. PMID 21436186